CLINICAL TRIAL: NCT05333887
Title: Moderators and Mediators of Behavioural Parent Training Outcomes for Children With Attention-deficit/Hyperactivity Disorder: Evaluating the Importance of Addressing Parent Psychopathology and Treatment Process Factors
Brief Title: Pilot Study of the Parental Friendship Coaching+ Program for Families of Children With Attention-deficit/Hyperactivity Disorder
Acronym: PFC+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amori Yee Mikami, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H21-00930
Record Dates: First submitted 2022-02-16; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: ADHD; Depression
Keywords: parent training; ADHD; friendship; mental health
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study attempts to modify a BPT program to be better suited to the needs of parents with mental health concerns. Modifications include ways to improve parent engagement and connection to the program. Parent engagement is often addressed by reducing practical barriers. All sessions are provided online, all strategies are presenting in a half-day group workshop, the remaining sessions only occur with 1-2 parents and are flexibly scheduled for the parent, a treatment menu is used to support easy tailoring of homework to family needs, and a general flexible approach is used. Programs also target parent connection via modifications to improve cognitions about treatment and ADHD, increase alliance, or increase treatment satisfaction. In the first two sessions barriers to treatment and unhelpful thoughts about treatment are discussed, the workshop is a group format, parents have the option to be put in pairs for social support, and they have a consistent therapist throughout the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFC+ (Experimental): In this condition, therapists instruct parents in ways to coach their children to display better friendship behaviours using skill teaching and home practice. The program includes 2 intake sessions, a group workshop where all strategies are reviewed, and 3 consultation sessions to work on implementing strategies with therapist support.
  Interventions: Behavioral: PFC+
- Waitlist (No Intervention): In this condition, parents are placed on a waitlist where they continue life as usual. After the waitlist they participate in the PFC+ program.

INTERVENTIONS:
Behavioral: PFC+ — Therapists instruct parents in ways to coach their children to display better friendship behaviours using skill teaching and home practice. The program includes 2 intake sessions, a group workshop where all strategies are reviewed, and 3 consultation sessions to work on implementing strategies with therapist support. Emphasis throughout the program is placed on parents' connection and engagement with the material and therapist.
  Arms: PFC+

SUMMARY:
Behavioural parent training (BPT) is a front-line treatment for children with attention-deficit/hyperactivity disorder (ADHD) that teaches parents how to support their child and manage behaviour. Parents of children with ADHD who have their own elevated ADHD/depressive symptoms may be less likely connect/engage and benefit from BPT. The current study modifies a BPT program that specifically addresses peer difficulties as these are common in children with ADHD. The goal of the modifications is to enhance the treatment process (how much parents connect and engage with the treatment) for parents with elevated ADHD/depressive symptoms. The Investigators will test whether this intervention increases parent engagement/connection to the program and whether it improves parenting behaviour.

DETAILED DESCRIPTION:
Study Purpose: The aim of this study is to conduct a pilot of PFC+ (a modified version of Parental Friendship Coaching), a BPT program for parents of children with ADHD and peer difficulties. Dr. Mikami created PFC and has conducted a randomized controlled trial comparing PFC to a psychoeducation/social support group. The investigators have modified PFC for parents with elevated ADHD and/or depressive symptoms to encourage engagement and connection with the program with the goal of improving eventual outcomes for these families. The reason why this modification was done is because parents with elevated ADHD and/or depressive symptoms typically do not benefit from BPT as much as parents without elevated symptoms. The current study examines the potential benefit of such modifications for these populations.

Hypothesis: The first hypothesis is that parents who participate in PFC+ will engage well with the program (attend, complete homework) and will report feeling connected to the program (satisfied with treatment, alliance with therapist, social support from parent peers). The second hypothesis is that participation in PFC+ will be associated with improvement in parenting related outcomes (parenting behaviour, parent stress, parent sense of competence), both over time and relative to a waitlist control condition.

Study Population: Participants will be families of children between the ages of 6-11. The parent will have elevated ADHD or depressive symptoms and will participate in the treatment and complete questionnaires and interviews. Children will have elevated ADHD symptoms and peer difficulties, and will complete questionnaires about the parent's parenting style. A co-parent will also be recruited, and can be anyone who can provide another perspective on the parent's parenting style (e.g., romantic partner, grandparent of the child); co-parents will complete questionnaires about the parent's parenting style.

Research Method: The investigators will recruit 48 parents to participate in the pilot of PFC+ and will use a crossover design so that all parents have the opportunity to participate in PFC+. In the eligibility screening, the parent will complete questionnaires about their symptoms and their child's symptoms to determine eligibility. At timepoint 1 (T1), all eligible families (parent, child, co-parent) will complete initial questionnaires to collect data about baseline functioning. Parents will be randomized to participate in PFC+ or a waitlist control condition (6 parents in each condition). PFC+ parents will then complete the treatment program over 5-6 weeks, while the waitlist parents will continue life as usual for 5-6 weeks. After PFC+ completes, all families will complete timepoint 2 (T2) questionnaires. Following this, crossover will occur, where parents in PFC+ will enter a naturalistic follow up, and parents previously in the waitlist condition will begin PFC+. Once treatment has finished (another 5-6 weeks), all families will complete timepoint 3 (T3) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Parents who participate in this study must meet the following criteria:

1. have a child (age 6-11) with elevated ADHD symptoms and peer difficulties;
2. have at minimum subclinical levels of depression and/or ADHD determined by self-report on symptom measures (parents with clinical levels are eligible);
3. be the primary parent involved with the child and their social life.

Exclusion Criteria:

Parents will be excluded if:

1. they cannot understand or speak English at a 9th grade level as they will be unable to participate in PFC+ (delivered in English) or complete questionnaires (reading/writing at the 9th grade level is not required as parents can be provided support in reading questionnaires and PFC+ content is delivered verbally);
2. they require alternative supports for more pressing mental health concerns (such that it would not be in their best interest to delay those other supports in order to participate in the current study), this might include schizophrenia, psychosis, a personality disorder, autism, intellectual disability, suicidal ideation, or self harm (they will be referred to alternative supports as needed);
3. they are participating in a different BPT program at the same time as they are projected to participate in PFC+;
4. if their 6-11 year old child has autism, pervasive developmental disorder, diagnosed or suspected intellectual disability, psychosis, or active suicidality (they will be referred to alternative supports as needed);
5. if their child does understand or speak English at the 1st grade level, as they will need to complete some questionnaires (research assistants will support children through questionnaires so reading at a 1st grade level is not required);
6. they do not have access to a computer, internet, and a private space to attend sessions (as the sessions are online, and a private space is needed to protect the confidentiality of other study participants).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Attendance (how many sessions did they attend) | The six possible sessions of the program in total, which occur over approximately 7 weeks
  - Descriptor: how many sessions did parents attend? This will be recorded after each session, and there are 6 possible sessions
Homework completion | The four possible sessions where homework is assigned, which occur over 4 weeks covering the last 4 sessions of the program
  - Descriptor: how often did parents complete their homework goals? Measured by the number of homework assignments that parents competed, out of four possible homework assignments
Time spent on material | The four possible sessions where homework is assigned, which occur over 4 weeks covering the last 4 sessions of the program
  - Descriptor: how many minutes did parents spend on program material outside of sessions. Measured by the total amount of minutes that parents spent on program material outside of session, over the entire program.
Early Working Alliance with Therapist (Working Alliance Inventory) | Measured in week 2 of the program (after session 2)
  - Descriptor: Therapeutic alliance
Post-Treatment Working Alliance with Therapist (Working Alliance Inventory) | Measured in week 7 (approximately one week after program completion)
  - Descriptor: Therapeutic Alliance
Group Social Support (Revised Working Alliance Inventory - Bond subscale) | Measured in week 7 (approximately one week after program completion)
  - Descriptor: Modified (WAI-SR) to report on bond between group members
Treatment Satisfaction | The six possible sessions of the program in total, which occur over approximately 7 weeks
  - Descriptor: how much did parents enjoy each session. Calculated as the average satisfaction with treatment, calculated as the mean of parent ratings of satisfaction obtained after each session.
Change in Parenting Behaviour After Program (Alabama Parenting Questionnaire) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in use of positive/negative parenting behaviours
Change in Parenting Behaviour at Follow-Up (Alabama Parenting Questionnaire) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in use of positive/negative parenting behaviours
Change in Parent Friendship Facilitation After Program (Friendship Facilitation Questionnaire) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in use of friendship facilitation skills
Change in Parent Friendship Facilitation at Follow-Up (Friendship Facilitation Questionnaire) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in use of friendship facilitation skills
Change in Parenting Stress After program (Parenting Stress Index - Short Form) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in parent stress levels
Change in Parenting Stress at Follow-Up (Parenting Stress Index - Short Form) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in parent stress levels
Change in Parenting Competence After Program (Parenting Sense of Competence Questionnaire) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in parent-reported levels of parenting competence
Change in Parenting Competence at Follow-Up (Parenting Sense of Competence Questionnaire) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in parent-reported levels of parenting competence

SECONDARY OUTCOMES:
Change in Child Peer Problems After Program (Strengths and Difficulties Questionnaire - Peer Problems Subscale) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in parent-reported child peer problems
Change in Child Peer Problems at Follow-Up (Strengths and Difficulties Questionnaire - Peer Problems Subscale) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in parent-reported child peer problems
Change in Child Quality of Play After Program (Quality of Play Questionnaire) | From baseline (week 0) to post-treatment (week 7; approximately one week after program completion)
  - Descriptor: Change in parent-reported child quality of play
Change in Child Quality of Play at Follow Up (Quality of Play Questionnaire) | From baseline (week 0) to follow-up (week 14; approximately seven weeks after program completion)
  - Descriptor: Change in parent-reported child quality of play

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Department of Psychology, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
In line with current best practices of psychological research, electronic de-identified data may be uploaded to a research repository or open science initiative for transparency and for possible future use. Any data shared through these initiatives will be uploaded in the form of a computer software file (e.g., SPSS) without any identifying information.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the main manuscript from the study is accepted, for 5 years.
Access Criteria: Investigator with doctoral degree in psychology or related field, or student being supervised by such an investigator.